CLINICAL TRIAL: NCT00004982
Title: Combination Iron Chelation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CHELATION (completed); 1R01DK055463-01 (NIH); NCT00004536 (obsolete NCT alias)
Record Dates: First submitted 2000-03-13; First posted 2000-03-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Iron Overload; Thalassemia
Keywords: chelation therapy; combination chemotherapy; iron poisoning; thalassemia; chelating agent; deferoxamine; drug screening /evaluation; therapy evaluation
MeSH Terms: conditions — Iron Overload; Thalassemia

INTERVENTIONS:
Drug: Combination Iron Chelation Therapy

SUMMARY:
Patients with beta-thalassemia (Cooley's Anemia) continue to suffer from the transfusion-induced iron overload due to the inadequacies of current iron-chelation therapy. Compliance with the use of the only FDA-approved drug for removing excess iron from patients (Desferal) continues to be a major problem despite convincing evidence that it markedly reduces morbidity and prolongs life. The full potential of iron-chelation therapy will not be realized until an orally-effective drug is available. This small trial is testing the premise that a combination of drugs as a new approach to iron chelation therapy may reduce side effects and increase efficacy. If both drugs can be given orally, there may be a better chance of finding a suitable alternative to Desferal. Several combinations of experimental iron chelating drugs are being used in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Iron overload

Exclusion Criteria:

* Overt cardiac disease

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-12; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University Medical College, New York, New York, United States